CLINICAL TRIAL: NCT05834010
Title: Feasibility Study of Using Fecal Microbiota Transplants (FMT) in Supportive Treatment of Anorexia Nervosa
Brief Title: Feasibility Study of Using Fecal Microbiota Transplants in Anorexia Nervosa
Acronym: ReBoot
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Collaborators: University of Copenhagen (Other); Odense University Hospital (Other); Psychiatric Center Ballerup (Other)
Responsible Party: Principal Investigator, Andreas Munk Petersen, Dr. MD pHD Clinical Associate Research Professor, Hvidovre University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H-22030034
Record Dates: First submitted 2023-03-18; First posted 2023-04-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Anorexia Nervosa; Microbiome Dysbiosis
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Intervention Model Description: 1 single FMT event either oral route or rectal. Sampling fecal matter and blood at baseline and 1 week after FMT.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- FMT (Experimental): rectal or oral route FMT
  Interventions: Biological: Fecal Microbiome Transplant

INTERVENTIONS:
Biological: Fecal Microbiome Transplant — Fecal matter from healthy age/sex matched established and screened donors, recruited from the Danish Blood-donor system
  Other Names: Fecal Matter Transplant

SUMMARY:
The investigators hypothesize that prolonged undernutrition in anorexia nervosa alters the microbiome to a different steady-state (dysbiotic) composition that sustains the disease, even after returning to normal diet. The investigators propose that transplanting a fully ecologically functioning GM from a healthy donor, through a FMT, can reboot the gut-brain-axis, ameliorate symptoms and improve clinical outcomes.

To approach this, in the challenging AN patient group, the investigators want to conduct a FMT feasibility/pilot study.

DETAILED DESCRIPTION:
Anorexia nervosa (AN) still carries the highest fatality rate of any psychiatric disease, and less than half of the patients recover, completely refractory to any treatment. The etiology remains unknown and evidence for treatment is lacking. We have an established collaboration bridging several disciplines and people in medicine, bioinformatics and biology with a focus on the pathological role of gut microbiome in the psychiatric disorder Anorexia nervosa. The GM in healthy people has been shown to affect weight gain, appetite and behavior through the gut-brain axis. We hypothesize that prolonged undernutrition in AN alters the microbiome to a different steady-state (dysbiotic) composition that sustains the disease, even after returning to normal diet. AN patients enter voluntarily into programs of therapeutic weight gain and reintroduction to normal food intake. The investigators propose that transplanting a fully ecologically functioning GM from a healthy donor, through a FMT, can reboot the gut-brain-axis, ameliorate symptoms and improve clinical outcomes. To approach this, in the challenging AN patient group, we want to conduct a FMT feasibility/pilot study. The investigators want approach the FMT intervention, with 20 AN patients in sequence before any attempt at more complex blinded /placebo clinical trials. The investigators will collect GM samples and clinical data from these patients and describe the altered composition and diversity of the AN-GM and how it changes with FMT.

Ultimately, the investigators aim to provide evidence that GM modulation with FMT can ameliorateclinical outcomes of AN. The investigators will investigate the feasibility of using FMT in supportive treatment of AN and by identifying specific bacterial and viral changes with FMT, we will lay the groundwork for randomized placebo-controlledstudies, to develop new GM interventions to complement current treatment of AN.

ELIGIBILITY:
Inclusion: Women referred to the participating specialized centers or by advertising who fulfill the of a diagnosis of Anorexia Nervosa according to the criteria as specified in the Diagnostic and Statistical Manual of Mental Disorders(DSM) version 5.

Exclusion:

Age <18 years. Known ongoing abuse of laxatives.

Antibiotic treatment within the last three months.

Probiotics within the last month

Inflammatory bowel disease, colorectal cancer or other known chronic bowel disorder

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2023-03-18 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of FMT in AN patients | 2 years
  The recruitment and compliance of 10-20 patients/year is feasible
Preferred route of FMT (questionnaire) | 2 years
  FMT is offered as a Capsule-treatment orally or as an enema-rectally

SECONDARY OUTCOMES:
A single FMT treatment can alter GM composition in AN patients short term | 2 yrs
  16S rRNA gene sequencing: Outcome: we expect GM to normalize towards the donor GM composition e.g higher diversity and composition of species, within the single patient and also compared to both healthy(NO-FMT) and AN(NO-FMT) controls.
A single FMT treatment can alter gut brain signaling in serum. might changes serum signal molecules related to appetite and metabolism with in same patien | 2 yrs
  measuring appetite related biomarkers: PYY might changes serum signal molecules related to appetite and metabolism with in same patient comparison, before and 1 week after FMT in a direction for higher appetite
A single FMT treatment can alter gut brain signaling in serum. might changes serum signal molecules related to appetite and metabolism with in same patien | 2 yrs
  measuring appetite related biomarkers: Leptin might changes serum signal molecules related to appetite and metabolism with in same patient comparison, before and 1 week after FMT in a direction for higher appetite
A single FMT treatment can alter gut brain signaling in serum. might changes serum signal molecules related to appetite and metabolism with in same patien | 2 yrs
  measuring appetite related biomarkers: Ghrelin,
A single FMT treatment can alter gut brain signaling in serum. might changes serum signal molecules related to appetite and metabolism with in same patien | 2 yrs
  measuring appetite related biomarkers: Insulin
A single FMT treatment can alter gut brain signaling in serum. might changes serum signal molecules related to appetite and metabolism with in same patien | 2 yrs
  measuring appetite related biomarkers: Glucagon
A single FMT treatment can alter gut brain signaling in serum. might changes serum signal molecules related to appetite and metabolism with in same patien | 2 yrs
  measuring appetite related biomarkers: GLP-1

OTHER OUTCOMES:
FMT questionnaires | 2 yrs
  With regards to the Pre and post FMT questionnaires we expect only to obtain patient narratives and guidance towards future designs since this is a feasibility study. We also hope to catch small self reported changes to "gut-feeling" in a positive direction. It is plausible that just one FMT might significantly lower discomfort as a result of changes to GM signaling. Again this serves only as a fesibility of using this type of questions in a future larger trial.

CONTACTS AND LOCATIONS:
Locations (3):
- Denmark (3):
  - Psychiatric Centre Ballerup, Ballerup Municipality, Denmark
  - Copenhagen University Hospital Hvidovre, Hvidovre, Denmark
  - Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Panah FM, Stoving RK, Sjogren M, Micali N, Maschek S, Reis KD, Mirsepasi-Lauridsen HC, Petersen AM, Nielsen DS, Helms M, Rasmussen MA, Barfod KK. Impact of a single fecal microbiome transplantation in adult women with anorexia nervosa: an open-label feasibility pilot trial. Nat Commun. 2026 Jan 14. doi: 10.1038/s41467-026-68455-8. Online ahead of print. PMID 41535289